CLINICAL TRIAL: NCT04645680
Title: Diet and Immune Effects Trial: DIET- A Randomized Double Blinded Dietary Intervention Study in Patients With Metastatic Melanoma Receiving Immunotherapy
Acronym: DIET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0158 (PA17-0104); NCI-2020-06112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0158 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-16; First posted 2020-11-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Unresectable Melanoma; Stage II Melanoma; Uveal Melanoma; Mucosal Melanoma; Unresectable Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded to their assigned diet throughout the intervention as will the investigators and research staff with the exception of the dietitian and the staff performing group assignment and data entry who will not have contact with participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (isocaloric high-fiber diet) (Experimental): Patients receive a whole foods diet that follows the recommended American Cancer Society guidelines but is higher in fiber for 11 weeks.
  Interventions: Other: Dietary Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (isocaloric diet) (Active Comparator): Patients receive a standard whole foods diet recommended by the American Cancer Society for 11 weeks.
  Interventions: Other: Dietary Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Dietary Intervention — Consume isocaloric whole foods diet higher in fiber
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (isocaloric high-fiber diet)
Other: Dietary Intervention — Whole foods diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm II (isocaloric diet)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This is a randomized, double-blind, fully controlled feeding study that will enroll melanoma patients starting standard-of-care ICB in three settings: adjuvant, neoadjuvant, and unresectable. Patients are randomized to the high fiber or healthy control diet. The goal of the study is to establish the effects of dietary intervention on the structure and function of the gut microbiome in patients with melanoma treated with SOC immunotherapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To establish the effects of dietary intervention on the structure and function of the gut microbiome.

SECONDARY OBJECTIVES:

1. Assess the effects of dietary intervention on gut metabolic output and systemic metabolism.
2. Assess the effects of dietary intervention on systemic and tumor immunity
3. Determine the safety (AEs) and tolerability (GSRS-IBS) of the dietary intervention
4. Assess the rate of immune related adverse events in patients on immunotherapy receiving dietary interventions
5. Determine the maximum daily fiber content that 70% of participants are able to tolerate
6. Assess the adherence to the dietary interventions as defined by 70% of calories consumed over the duration of the study being derived from provided diets (as measured by food records)
7. Assess the effects of dietary interventions on quality of life and other patient reported outcomes (PROs)

EXPLORATORY OBJECTIVES:

1. Assess the association of dietary interventions with clinical outcomes (objective response rate [ORR] and progression-free survival [PFS] rate in unresectable cohort and recurrence rate [RR] in adjuvant cohort).
2. Explore predictors of biological response to dietary interventions.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (ISOCALORIC HIGH-FIBER DIET): Patients receive a whole foods diet that follows the recommended American Cancer Society guidelines but is higher in fiber for 11 weeks.

ARM II (ISOCALORIC CONTROL DIET): Patients receive a standard whole foods diet of recommended by the American Cancer Society for 11 weeks.

After completion of study, patients are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Body mass index (BMI) 18.5-40 kg/m^2
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. English-speaking
5. Self-reported willingness to exclusively eat the provided diets
6. Self-reported willingness to comply with scheduled visits, undergo venipuncture, and provide stool samples
7. Cohort-specific:

   * 1 Adjuvant Melanoma: i. Resected Stage II-IV melanoma with planned initiation of adjuvant anti-PD1 +/- anti-CTLA4 or anti-LAG3
   * 2 Unresectable Melanoma: i. Histologically confirmed unresectable stage III or Stage IV melanoma with planned initiation of standard of care anti-PD1 +/- CTLA4 or anti-PD1 +/- LAG3 immunotherapy and no prior immunotherapy in the metastatic setting.
   * 3 Neoadjuvant Melanoma: i. Histologically confirmed stage III/IV melanoma with planned initiation of neoadjuvant anti-PD1 +/- anti-CTLA4 or anti-LAG3 1. Participants must have archival tissue block available or be willing to undergo a newly-obtained core needle or incisional biopsy at baseline. Fine needle aspiration is not acceptable.
   * 4 Unresectable RCC: i. Unresectable clear-cell renal cell carcinoma with planned initiation of standard of care anti-PD1 +/- anti-CTLA4 immunotherapy

Exclusion Criteria:

1. History of >= grade II colitis or diarrhea on immunotherapy or any ongoing colitis or diarrhea of any grade
2. Unresolved >= grade III immune-related adverse event on immunotherapy (other than endocrinopathy requiring hormone replacement)
3. History of active inflammatory bowel disease or major gastrointestinal surgery (not including appendectomy or cholecystectomy) within 3 months of enrollment or any history of total colectomy, or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, i.e. restrictive procedures such as banding, are permitted).
4. Medical contraindications to intervention diet as determined by the treating physician
5. Self-reported major dietary restrictions related to the intervention
6. Diagnosis of diabetes mellitus type I or type II that requires medical treatment or random glucose > 200 mg/dL
7. Antibiotic use within 21 days of planned start of equilibration diet (self-reported and/or noted by the treating physician)
8. Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study intervention administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
9. Regularly taking probiotics, fiber supplements, or any other medication or supplement that could affect study outcome as determined by the principal investigator and unable/unwilling to discontinue for the purpose of the study. These agents must be discontinued at least 14 days prior to start of diet
10. Currently consuming an average estimated daily fiber intake exceeding 20 grams based on the results of the preliminary dietary assessment; vegetarian or vegan
11. Current smoker or heavy drinker (defined as > 14 drinks per week) or current self reported illicit drug use
12. Uncontrolled concurrent illness or infection or psychiatric illness/social situations that would limit compliance with study requirements
13. Unable or unwilling to undergo study procedures
14. Plan for travel during the study that would preclude adherence to prescribed diets
15. Cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in the gut microbiome | Baseline up to 11 weeks
  Changes of alpha-diversity (e.g., Shannon index) and abundance/relative abundance of different taxon levels (e.g., genus, family), from baseline to end of intervention, will be estimated. The outcomes will be compared. between two arms using t-test or Mann-Whitney test. Linear mixed effects models will be used for assessing the longitudinal data. Similarity in microbiome community structure will be assessed using principal coordinate analysis (PCoA) and compared using multivariate analysis of variance (MANOVA).

SECONDARY OUTCOMES:
Change in systemic and tumor immunity | Up to 12 weeks
  Percent change in CD8 T cells using flow cytometry will be compared between two arms using t-test or Mann-Whitney test. Pearson or Spearman correlation coefficient will be used to assess the correlation between the outcome at baseline and end of intervention.
Change in metabolic profile | Baseline up to 11 weeks
  Change in relative concentration (ion intensity determined as area under the curve) measured by mass spectrometry-based analysis of blood and fecal specimens from baseline to end of intervention will be compared between two arms using t-test or Mann-Whitney test.
Change in quality of life (QOL) | Baseline up to 11 weeks
  Change in quality of life between baseline and end of intervention using a validated, 30 question scoring instrument (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Each question is scored in from 1 ("not at all") to 4 ("very much") in a Likert format. Linear mixed effects models will be used for assessing the longitudinal data. Pearson or Spearman correlation coefficient will be used to assess the correlation between measures for quality of life at baseline and end of intervention.
Incidence of adverse events | Up to 12 weeks
  AEs attributed to diet as well as immune-related adverse events (irAEs) attributed to immunotherapy will be assessed using frequency counts and percentages.
Symptom profile | Up to 12-week follow-up
  To assess gastrointestinal symptoms related to the dietary interventions, the GSRS-IBS will be used. The GSRS-IBS is a 13-item validated instrument with subscales for each item ranging from 0 ("no discomfort at all") to 7 ("very severe discomfort"). The gastrointestinal symptoms (GSRS-IBS) will be summarized using frequency counts and percentages.

OTHER OUTCOMES:
Objective response rate (ORR) (unresectable cohort) | At 12-week follow-up
  Response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The ORR will be estimated along with 95% confidence interval, and compared between two diet groups using Chi-squared test or Fisher's exact test as appropriate.
Progression-free survival (PFS) (unresectable cohort) | Up to 12-week follow-up
  Response will be assessed by RECIST 1.1. PFS will be assessed using Kaplan-Meier method and compared between two diet groups using log-rank test.
Recurrence rate (RR) (adjuvant cohort) | Up to 12-week follow-up
  Response will be assessed by RECIST 1.1. The RR will be estimated along with 95% confidence interval, and compared between two diet groups using Chi-squared test or Fisher's exact test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Baruch, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Farias RM, Jiang Y, Levy EJ, Hwang C, Wang J, Burton EM, Cohen L, Ajami N, Wargo JA, Daniel CR, McQuade JL. Diet and Immune Effects Trial (DIET)- a randomized, double-blinded dietary intervention study in patients with melanoma receiving immunotherapy. BMC Cancer. 2024 Dec 4;24(1):1493. doi: 10.1186/s12885-024-13234-1. PMID 39633321
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04645680/ICF_000.pdf